CLINICAL TRIAL: NCT05190380
Title: COMPARATIVE EFFECTS OF HIGH AND LOW INTENSITY PROGRESSIVE RESISTED EXERCISES ON PAIN, RANGE OF MOTION AND FUNCTIONAL DISABILITY IN KNEE OSTEOARTHRITIS PATIENTS WITH SARCOPENIA: A RANDOMIZED CONTROLLED TRIAL
Brief Title: HIGH AND LOW INTENSITY PROGRESSIVE RESISTED EXERCISES ON PAIN, RANGE OF MOTION AND FUNCTIONAL DISABILITY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Saiqa Kanwal, COMPARATIVE EFFECTS OF HIGH AND LOW INTENSITY PROGRESSIVE RESISTED EXERCISES ON PAIN, RANGE OF MOTION AND FUNCTIONAL DISABILITY IN KNEE OSTEOARTHRITIS PATIENTS WITH SARCOPENIA: A RANDOMIZED CONTROLLED TRIAL, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/981/2021
Record Dates: First submitted 2021-12-30; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Osteo Arthritis Knee; Sarcopenia
Keywords: osteoarthritis; Sarcopenia
MeSH Terms: conditions — Sarcopenia; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity (Experimental): Intervention: Leg presses, knee extension, hip adduction and hip abduction exercises will be performed by patients. There will be a warm up sets for 1 repetition maximum with 2 min gap between both sets (leg press + knee extension exercises) (hip abduction and hip adduction) patients will ask to perform.Routine physical therapy including TENS, Hot pack and Deep friction massage along with high intensity exercises will also be delivered along with Muscle Energy Technique. Experimental:High intensity will be treated with high intensity exercises in such a way that
  1st and 2nd week; resistance training will be of 50% 1RM with 4 sets of 10 repetitions.
  3rd and 4th week: resistance training will be of 70% 1RM with 4 sets of 10 repetitions.
  5th and 6th week: the training will be of 80% 1RM with 4 sets of 10 repetitions
  Last 4 sessions will be:
  7th and 8th week: resistance training will be of 80% 1RM with 5 sets of 10 repetitions.
  Interventions: Other: HIGH INTENSITY PROGRESSIVE RESISTED EXERCISE
- Low intensity (Experimental): Intervention: Leg presses, knee extension, hip adduction and hip abduction exercises will be performed by patients. There will be a warm up sets for 1 repetition maximum with 2 min gap between both sets (leg press + knee extension exercises) (hip abduction and hip adduction) patients will ask to perform.Routine physical therapy including TENS, Hot pack and Deep friction massage along with Low intensity exercises will also be delivered along with Muscle Energy Technique. Experimental:Low intensity Group B will be treated with low intensity exercise in such a way that,
  1st and 2nd week; Resistance training will be of 20% 1RM with 4 sets of 15 reps 3rd and 4th week Resistance training will be of 30% 1RM with 4 sets of 15 reps 5th and 6th week: the training will be of 40% 1RM with 4 sets of 15 reps
  Last session will be:
  7th and 8th week; Training of 40% 1RM with 5 sets of 15 reps
  Interventions: Other: LOW INTENSITY PROGRESSIVE RESISTED EXERCISE

INTERVENTIONS:
Other: HIGH INTENSITY PROGRESSIVE RESISTED EXERCISE — Intervention:Leg presses, knee extension, hip adduction and hip abduction exercises will be performed by patients. There will be a warm up sets for 1 repetition maximum with 2 min gap between both sets (leg press + knee extension exercises) (hip abduction and hip adduction) patients will ask to perform.
  Both groups will receive routine physical therapy (Tens, Hot pack, Deep friction massage) in addition with experimental interventions
  Arms: High intensity
Other: LOW INTENSITY PROGRESSIVE RESISTED EXERCISE — Intervention:Leg presses, knee extension, hip adduction and hip abduction exercises will be performed by patients. There will be a warm up sets for 1 repetition maximum with 2 min gap between both sets (leg press + knee extension exercises) (hip abduction and hip adduction) patients will ask to perform.
  Both groups will receive routine physical therapy (Tens, Hot pack, Deep friction massage) in addition with experimental interventions
  Arms: Low intensity

SUMMARY:
The study will be randomized controlled trial. This study will be conducted in University of Lahore Teaching Hospital, Lahore, Pakistan. A sample size of 84 will be randomly allocated into two experimental groups, (42 participants in each group), by computer generated random number list. The participants,randomly allocated to the experimental group A, will receive high intensity resisted exercises ,in addition with routine physical therapy as TENS (transcutaneous electrical nerve stimulator), Hot pack, Deep friction massage Each session will be of 35-45 minutes with 5 minutes warm up, 35 minutes for training session and lastly 5 minutes for cool down

• Participants in experimental group B, will receive Low intensity resisted exercises in addition with routine physical therapy

DETAILED DESCRIPTION:
Recruitment: Participants will be recruited and referred by orthopedic doctor, University of Lahore Teaching Hospital to Physical Therapy Department. The study will be randomized controlled trial. This study will be conducted in University of Lahore Teaching Hospital, Lahore, Pakistan. A sample size of 84 will be randomly allocated into two experimental groups, (42 participants in each group), by computer generated random number list. The participants,randomly allocated to the experimental group A, will receive high intensity resisted exercises ,in addition with routine physical therapy as TENS, Hot pack, Deep friction massage

* Participants in experimental group B, Low intensity resisted exercises in addition with routine physical therapy
* Both experimental groups will receive sixteen treatment sessions and those will be given over a period of eight weeks (2 sessions per week, each session of 35-45 minutes with 5 minutes warm up and lastly 5 minutes for cool down in both groups.
* Outcome measure will be taken by assessor at baseline, and at the end of 8th week (at the end of last treatment session) through Numeric pain rating scale and KOOS
* Randomization and Allocation: Afterwards, participants confirming the eligibility criteria will be randomly allocated, through computer generated random number list , into two experimental groups (Group A, Group B).
* Blindness: Study will be single, assessor blinded and an independent investigator will perform randomization and will inform the patients and therapist about the allocation.
* Intervention: Leg presses, knee extension, hip adduction and hip abduction exercises will be performed by patients. There will be a warm up sets for 1 repetition maximum with 2 min gap between both sets (leg press + knee extension exercises) (hip abduction and hip adduction) patients will ask to perform.
* Duration: Sixteen treatment sessions will be given over a period of eight weeks (2 sessions per week, each session of 35-45 minutes).
* Outcome Variables and Measures

  1. Pain (Numeric pain rating scale)
  2. Functional disability (KOOS)
  3. ROM (Universal Goniometer)
* Outcome measures will be taken at baseline and at the end of last treatment session i.e. 8th week. Collected data will be than analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Age range between 35-65 years
* Diagnosed osteoarthritis patients of grade I to III according to kellgren & Lawrence on X-ray (diagnosed by orthopedic specialist)
* Diagnosed patients with sarcopenia according to SARC-F questionnaire. (diagnosed by orthopedic specialist)

Exclusion Criteria:

* Patients with history of trauma like RTA(road traffic accident)

  , fall history and other loading injuries, patellar fracture or dislocation.
* Patients with history of surgery (meniscal reconstruction, TKR(total knee replacement) or Partial Knee Replacement etc.)
* Patients with severe patellofemoral osteoarthritis.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-07-08 (Estimated); Study Completion 2022-07-18 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 8 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain
Knee injury and Osteoarthritis Outcome Score (KOOS) | 8 weeks
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. The KOOS evaluates both short-term and long-term consequences of knee injury. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL)
Range of motion | 8 weeks
  Range of motion is the extent of movement of a joint, measured in degrees of a circle. Universal goniometer (UG) will be used to evaluate range of motion (ROM)

CONTACTS AND LOCATIONS:
Overall Officials: Saiqa Kanwal, MS-MSK*, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Pickering ME, Chapurlat R. Where Two Common Conditions of Aging Meet: Osteoarthritis and Sarcopenia. Calcif Tissue Int. 2020 Sep;107(3):203-211. doi: 10.1007/s00223-020-00703-5. Epub 2020 May 18. PMID 32424600
- [Background] Bade MJ, Struessel T, Dayton M, Foran J, Kim RH, Miner T, Wolfe P, Kohrt WM, Dennis D, Stevens-Lapsley JE. Early High-Intensity Versus Low-Intensity Rehabilitation After Total Knee Arthroplasty: A Randomized Controlled Trial. Arthritis Care Res (Hoboken). 2017 Sep;69(9):1360-1368. doi: 10.1002/acr.23139. Epub 2017 Aug 13. PMID 27813347
- [Background] Messier SP, Mihalko SL, Beavers DP, Nicklas BJ, DeVita P, Carr JJ, Hunter DJ, Lyles M, Guermazi A, Bennell KL, Loeser RF. Effect of High-Intensity Strength Training on Knee Pain and Knee Joint Compressive Forces Among Adults With Knee Osteoarthritis: The START Randomized Clinical Trial. JAMA. 2021 Feb 16;325(7):646-657. doi: 10.1001/jama.2021.0411. PMID 33591346
- [Background] Liao CD, Chiu YS, Ku JW, Huang SW, Liou TH. Effects of Elastic Resistance Exercise on Postoperative Outcomes Linked to the ICF Core Sets for Osteoarthritis after Total Knee Replacement in Overweight and Obese Older Women with Sarcopenia Risk: A Randomized Controlled Trial. J Clin Med. 2020 Jul 11;9(7):2194. doi: 10.3390/jcm9072194. PMID 32664548
- [Background] Thorstensson CA, Roos EM, Petersson IF, Ekdahl C. Six-week high-intensity exercise program for middle-aged patients with knee osteoarthritis: a randomized controlled trial [ISRCTN20244858]. BMC Musculoskelet Disord. 2005 May 30;6:27. doi: 10.1186/1471-2474-6-27. PMID 15924620
- [Background] Shorter E, Sannicandro AJ, Poulet B, Goljanek-Whysall K. Skeletal Muscle Wasting and Its Relationship With Osteoarthritis: a Mini-Review of Mechanisms and Current Interventions. Curr Rheumatol Rep. 2019 Jun 15;21(8):40. doi: 10.1007/s11926-019-0839-4. PMID 31203463